CLINICAL TRIAL: NCT00820313
Title: Coronary Events, Risk Factors, and Quality of Life in Men and Women Enrolled in Intensive Lifestyle Interventions - A Prospective Evaluation of Health Services Outcomes and Emerging Cardiovascular Disease Biomarkers
Brief Title: A Prospective Evaluation of Health Services Outcomes and Emerging Cardiovascular Disease Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Preventive Medicine Research Institute (Other)
Responsible Party: Dean Ornish, MD, Preventive Medicine Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPMC-26.096SLH; W81XHW-06-1-0565
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Heart Disease; Biomarkers of Cardiovascular Disease
Keywords: Coronary Heart Disease; Biomarkers of Cardiovascular Disease; Health Related Quality of Life; Diabetes; Diet
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Intervention (Other): Comprehensive lifestyle intervention for reversal of heart disease
  Interventions: Behavioral: Dr. Dean Ornish Program for Reversing Heart Disease

INTERVENTIONS:
Behavioral: Dr. Dean Ornish Program for Reversing Heart Disease — Exercise: At least 3 hours of aerobic exercise per week, 30 minutes per session. Additionally, patients are asked to perform a minimum of 2 strength training sessions per week.
  Stress Management: Integrates stretching, relaxation, breathing techniques, meditation and guided imagery. Patients are asked to practice these techniques at least 1 hour per day.
  Diet: Approximately 10% daily calories from fat, 15% protein and 75% complex carbohydrates (low-fat, whole foods, primarily plant-based).
  Group Support: Weekly group support sessions provide social support to help patients adhere to and sustain the lifestyle-change program.

SUMMARY:
The primary aim of the proposed research is to examine the relationship of lifestyle changes to new dietary, biomedical, and cellular parameters among new enrollees entering the "Dr. Dean Ornish Program for Reversing Heart Disease program" at 5 selected sites. Specifically, the investigators will add assessments of emerging cardiac risk factors (e.g., high sensitivity C-reactive protein [hsCRP], fibrinogen, lipoprotein(a) [Lp(a)], small, dense LDL, apolipoprotein B [apoB], apolipoprotein A-I [apo A1], the apoB/apoA1 ratio, homocysteine [Hcy], B-type natriuretic peptide [BNP], oxidized LDL, fasting insulin and waist-to-hip ratio [WHR]), protective and pathogenic dietary markers (e.g., folate, carotenoids, trans fatty acids), and measures of social support and cognitive functioning to the already existing assessment variables in the Multisite Cardiac Lifestyle Intervention Program (MCLIP).

Hypothesis 1: Participation in the lifestyle program will not only be associated with favorable changes in standard coronary risk factors and quality of life, but also with improvements in emerging cardiac risk factors [hsCRP, Hcy, BNP, fibrinogen, Lp(a), small, dense LDL, apoB, apoA1, oxidized LDL, fasting insulin, and abdominal obesity] and psychosocial well-being (i.e., social support, and cognitive functioning).

Hypothesis 2: High intake of emerging protective dietary factors and low intake of emerging pathogenic dietary factors will be associated with improvements in both standard and emerging cardiac risk factors (e.g. Hcy, oxidized LDL).

Hypothesis 3: Degree of adherence to the lifestyle change program will be associated with differential improvement in standard coronary risk factors, emerging risk factors, cellular aging, and psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients included those who had a diagnosis of coronary heart disease (CHD) from their physician or health plan, a diagnosis of diabetes, or at least 3 additional cardiac risk factors.
* A diagnosis of CHD included:

  * having diagnosed CHD based on non-invasive testing such as exercise testing, nuclear imaging, echocardiogram or other test that clearly demonstrates ischemia
  * cardiac catheterization demonstrating CHD
  * eligibility for bypass surgery/PTCA and seeking a clinical alternative
  * coronary bypass surgery
  * PTCA/stent
  * myocardial infarction.
* Type I or Type II diabetics were eligible for the program.
* For a participant to be included as a high-risk factor participant, the participant must have either a family history of premature CHD (1st-degree relative (male<55; female <65) with MI or sudden cardiac death) or be a male aged > 45 or a female aged > 55.
* In addition, there must be at least two additional cardiovascular risk factors, including:

  * current cigarette smoking (within the past 5 years)
  * hypertension: BP > 140/90 mm Hg or on antihypertensive medication,
  * low HDL-C: <35 mg/dl or on medications for lipid therapy
  * elevated apolipoprotein(a): >30 mg/dl or on medications for elevated lipids
  * high total cholesterol: > 240 or on medications for elevated lipids
  * high LDL-C: >160 or on medications for elevated lipids
  * high sensitivity C-Reactive Protein: > 3 mg/dl and < 10 mg/dl
  * obesity: BMI > 30
  * Insulin Resistant State (Metabolic Syndrome X

Exclusion Criteria:

* Exclusion criteria included:

  * ischemic left main CHD, with an obstruction greater than 50%
  * significant (>70%) proximal left anterior descending artery disease and proximal left circumflex artery disease and an ejection fraction less than 50%, *unstable angina
  * hypotensive response to exercise (> 20mm Hg drop in systolic BP)
  * history of exercise induced ventricular tachycardia or 3rd degree heart block without evidence of current stability
  * CABG surgery within 4 weeks, unless approved by medical director
  * MI within one month, unless approved by medical director\
  * HF, with functional limitation and unresponsive to medications
  * current tobacco user not concurrently enrolled in a smoking cessation program with 2-month history of smoking cessation
  * uncontrolled malignant ventricular arrhythmia despite medications and/or implantable cardiac defibrillator (ICD), unless approved by medical director, resides beyond a one-hour commute to the Program site, unless approved by Team, *history of substance abuse disorder (inc. ETOH) without documentation of a minimum one year of abstinence
  * history of a significant psychiatric disorder without documentation of minimum one-year stability
  * impaired cognitive function, such as dementia or delirium
  * English language literacy unless Program site can accommodate
  * non-ambulatory
  * uncooperative spouse or life partner, defined as obstructive in attitude or behavior
  * the patient is deemed to be potentially disruptive to group setting by the screening team.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of Cardiovascular Disease | Baseline Assessment, 3 month Follow-up Assessment, 12 month Follow-up Assessment

SECONDARY OUTCOMES:
Dietary Intake | Baseline Assessment, 3 month Follow-up Assessment, 12 month Follow-up Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kersh, MD, FACC, Principal Investigator — St. Luke's Hospital/California Pacific Cardiovascular Medical Group, Inc; Dean Ornish, MD, Principal Investigator — Preventive Medicine Research Institute; Gerdi Weidner, PhD, Principal Investigator — Preventive Medicine Research Institute; Nita Chainani-Wu, DMD, MS, PhD, Study Director — Preventive Medicine Research Institute
Locations (1):
- Preventive Medicine Research Institute, Sausalito, California, United States

REFERENCES:
- [Background] Govil SR, Weidner G, Merritt-Worden T, Ornish D. Socioeconomic status and improvements in lifestyle, coronary risk factors, and quality of life: the Multisite Cardiac Lifestyle Intervention Program. Am J Public Health. 2009 Jul;99(7):1263-70. doi: 10.2105/AJPH.2007.132852. Epub 2008 Oct 15. PMID 18923113
- [Background] Pischke CR, Scherwitz L, Weidner G, Ornish D. Long-term effects of lifestyle changes on well-being and cardiac variables among coronary heart disease patients. Health Psychol. 2008 Sep;27(5):584-92. doi: 10.1037/0278-6133.27.5.584. PMID 18823185
- [Background] Schulz U, Pischke CR, Weidner G, Daubenmier J, Elliot-Eller M, Scherwitz L, Bullinger M, Ornish D. Social support group attendance is related to blood pressure, health behaviours, and quality of life in the Multicenter Lifestyle Demonstration Project. Psychol Health Med. 2008 Aug;13(4):423-37. doi: 10.1080/13548500701660442. PMID 18825581
- [Background] Frattaroli J, Weidner G, Merritt-Worden TA, Frenda S, Ornish D. Angina pectoris and atherosclerotic risk factors in the multisite cardiac lifestyle intervention program. Am J Cardiol. 2008 Apr 1;101(7):911-8. doi: 10.1016/j.amjcard.2007.11.039. Epub 2008 Jan 28. PMID 18359307
- [Background] Pischke CR, Weidner G, Elliott-Eller M, Ornish D. Lifestyle changes and clinical profile in coronary heart disease patients with an ejection fraction of <or=40% or >40% in the Multicenter Lifestyle Demonstration Project. Eur J Heart Fail. 2007 Sep;9(9):928-34. doi: 10.1016/j.ejheart.2007.05.009. Epub 2007 Jun 14. PMID 17572148
- [Background] Daubenmier JJ, Weidner G, Sumner MD, Mendell N, Merritt-Worden T, Studley J, Ornish D. The contribution of changes in diet, exercise, and stress management to changes in coronary risk in women and men in the multisite cardiac lifestyle intervention program. Ann Behav Med. 2007 Feb;33(1):57-68. doi: 10.1207/s15324796abm3301_7. PMID 17291171
- [Background] Ornish D, Weidner G, Fair WR, Marlin R, Pettengill EB, Raisin CJ, Dunn-Emke S, Crutchfield L, Jacobs FN, Barnard RJ, Aronson WJ, McCormac P, McKnight DJ, Fein JD, Dnistrian AM, Weinstein J, Ngo TH, Mendell NR, Carroll PR. Intensive lifestyle changes may affect the progression of prostate cancer. J Urol. 2005 Sep;174(3):1065-9; discussion 1069-70. doi: 10.1097/01.ju.0000169487.49018.73. PMID 16094059
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- See also: Preventive Medicine Research Institute website homepage — http://www.pmri.org/